CLINICAL TRIAL: NCT06281444
Title: Effectiveness of the Effect of Radial Extracorporeal Shock Wave Therapy in Addition to Exercise on Pain, Functionality and Walking Distance in Patients With Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Effectiveness of Radial Extracorporeal Shock Wave Therapy in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Birkan Sonel Tur, Clinical Professor (Physical Medicine and Rehabilitation), Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: i01-30-24
Record Dates: First submitted 2024-02-07; First posted 2024-02-28 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Extracorporeal shock wave therapy (ESWT); Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: Patients who accepted to participate in the study by meeting the criteria will be randomly divided into two groups as the first group treatment ESWT + exercise, the second group sham ESWT + exercise.
Who Masked: Participant
Masking Description: Patients who meet the study conditions and agree to participate in this study will not know whether they are in the first group or the second group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT group (Active Comparator): The participants in this group will be applied with ESWT plus a home-based exercise program.
  Interventions: Device: ESWT
- Sham-ESWT group (Sham Comparator): The participants in this group will be applied with sham-ESWT plus a home-based exercise program.
  Interventions: Device: Sham-ESWT

INTERVENTIONS:
Device: ESWT — All patients in both groups will be applied with a home-based exercise program around for 30-minutes per day for four weeks. The exercises that mentioned in the research content are knee range of motion and strengthening exercises for the knee. It will be checked by phone on a weekly basis. Also, each patient in group 1 will receive shockwaves of continuous frequency and intensity (1000 shocks, 2.0 to 3.0 bar,10 Hz and 0.08-0.25mJ/mm2 energy range), while the second group of patients will receive sham-ESWT.
  ESWT application will be applied to the medial part of the knee area on the side where the pain is described, or at the patellofemoral and tibiofemoral borders of the affected knee, and will be given in four sessions in total once a week.
  Arms: ESWT group
Device: Sham-ESWT — Sham ESWT application will be set to 1000 pulses, 2-3 bar pressure, 10 Hz frequency and 0 mJ/mm2 energy to be sham.
  Arms: Sham-ESWT group

SUMMARY:
Osteoarthritis (OA) is a degenerative joint disease characterized by unsuccessful repair of joint damage resulting from stresses in any of the synovial joint tissues. Symptoms include pain (initially only after movement), joint stiffness, limitation of joint movement, feeling of insecurity in the joint, and difficulty walking. The diagnosis of knee osteoarthritis can be easily made with a detailed history and a comprehensive physical examination. Radiographic examinations are used to support clinical findings and exclude other possible pathologies. The main purpose of treating knee osteoarthritis is to reduce pain and make daily life easier. Since there is no standard treatment method, the patient's treatment must be individualized by taking into account age, comorbidity, severity of the clinical picture, patient preferences and cost of treatment. Conservative treatment includes pharmacological and non-pharmacological treatment, and the optimal treatment should be applied as a combination of these two methods. Patient education, lifestyle modification, exercise, different physical therapy modalities (TENS, Interferential current, ESWT...), acupuncture are some non-pharmacological methods.

Extracorporeal shock wave therapy (ESWT), which is considered within the scope of conservative treatment, started in the seventies with the practice of breaking ureteric stones and has become one of the physical therapy modalities used in the treatment of various musculoskeletal diseases. Considering the historical development of ESWT, it has started to be used as a therapeutic modality in the treatment of knee osteoarthritis in recent years. The process, which started with animal experiments, continued with human studies, and evidence is presented that ESWT reduces knee pain and contributes to functionality. It is noteworthy that there are few studies and their short follow-up periods. In the light of these studies, it was planned to investigate the effectiveness of ESWT treatment, which will be applied together with exercise, on pain, functionality and walking distance in individuals diagnosed with knee osteoarthritis, in comparison with the control group receiving sham ESWT.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled trial. Eligible patients who meet the inclusion criteria, will be invited to the study.

Patients who accepted to participate in the study by meeting the criteria will be randomly divided into two groups as the first group treatment ESWT + exercise, the second group sham ESWT + exercise. Computer-aided software will be used to assign patients to treatment groups.

The following evaluations will be made: Visual Analog Scale (VAS), Patient Global Assessment (PGA), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and 6-minute walk test (6MWT).

VAS is widely used in the assessment of pain. In the present study, pain was assessed in three conditions: at rest, during movement, and at night.

PGA is an instrument used in clinical settings to capture the patient's subjective appraisal of overall health and disease-related well-being, serving as a concise indicator of disease activity.

WOMAC is widely used to evaluate the functional status of patients with knee osteoarthritis. High WOMAC values indicate increased pain and stiffness/stiffness, and impaired physical function.

6MWT will be done by the physician in the marked corridor of 30 meters in our clinic. At the end of 6 minutes, the total distance they walked will be determined and recorded in meters.

The exercises to be applied to each group are knee range of motion and strengthening exercises for the knee. It will be checked by phone on a weekly basis.

The first group will receive ESWT and exercise therapy. ESWT application will be given to the medial part of the knee region on the side where the pain is described, on the patellofemoral and tibiofemoral joint lines and once a week in a total of four sessions.

The second group will receive sham ESWT and exercise therapy. Sham ESWT application will be given to the medial part of the knee region on the side where the pain is described, on the patellofemoral and tibiofemoral joint lines and once a week in a total of four sessions.

Before starting the 4-session treatment program, at the end of the treatment program and at the twelfth, twenty-fourth weeks from the beginning of the treatment, the scales and tests under the heading of evaluations will be administered.

The sample calculation was made on the effect size. When the effect size of the difference between the two treatment groups in terms of change in VAS is taken as 0.8, when the sample is calculated using the Mann-Whitney U test with a significance level of 0.05 and a power of 0.85, the sample study is 36 patients per group and a total of 72 patients in total was found to be sufficient.

ELIGIBILITY:
Inclusion Criteria:

* Being over 50-85 years old.
* Diagnosis of knee osteoarthritis according to ACR clinical/radiological diagnostic criteria
* Stage 2 and above according to Kellgren Lawrence (K-L)
* Completion of Informed Signed Consent Form

Exclusion Criteria:

* Gait disorders due to orthopedic or neuromuscular disease
* Participation in a structured physical rehabilitation program in the last 12 months before the study
* Those who have had an intra-articular injection of the knee in the last 6 months
* History of lower extremity surgery
* Those with mechanical instability in the knee, a history of infection, malignancy
* Inflammatory rheumatic diseases (rheumatoid arthritis, spondyloarthritis etc.)
* A medical diagnosis or self-reported cognitive impairment
* Presence of progressive cancer AND/OR other diseases that impair general condition
* Situations where ESWT application is contraindicated
* Having previously received ESWT treatment
* Patients with hip and/or ankle pathology

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Change in pain [by using the Visual Analogue Scale(VAS)] | Up to 24 weeks
  It was defined as the change in pain (VAS) felt after 4 sessions of ESWT treatment from baseline.
  Visual Analog Scale (VAS): Vas is widely used in pain assessment. The numbers 0 and 10 are written at both ends of a 10 cm line. 0 = I have no pain 10 = means I have unbearable pain. The pain level increases from 0 to 10. The patient is asked to indicate which point on this chart is most appropriate for his/her situation. The location marked by the patient will be evaluated by measuring its distance from point 0.

SECONDARY OUTCOMES:
Change from baseline in functionality and walking distance | Up to 24 weeks
  Change from baseline in functionality (WOMAC) and walking distance (6-minute walk test)
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): WOMAC is widely used to evaluate the functionality status in patients with knee osteoarthritis.
  High WOMAC values indicate increased pain and stiffness and deterioration in physical function.
  The form consists of three subheadings (pain, stiffness, physical function) and 24 questions.
  The pain subheading is questioned with 5 questions, and the stiffness subheading is questioned with 2 questions. In the physical function evaluation, 17 activities are questioned.
  Scoring of the items is done according to the Likert scale. The degree of pain and strain is indicated by giving points from 0 to 4 on the Likert scale.
Change from baseline in walking distance | Up to 24 weeks
  Change from baseline in walking distance (6-minute walk test)
  6-minute walk test: It will be performed by the physician in the 30-meter marked corridor in our clinic. Patients will be asked to rest for at least 10 minutes before starting the test.
  Patients will be asked to walk as far as they can in the corridor for 6 minutes at their own pace.
  At the end of 6 minutes, the total distance walked will be determined and recorded in meters.
Patient Global Assesment (PGA) [by using the VAS] | Up to 24 weeks
  It was defined as the change in PGA felt after 4 sessions of ESWT treatment from baseline.
  The Patient Global Assessment (PGA) is a measure used in clinical research and routine practice to capture the patient's subjective evaluation of their overall health status and disease-related well-being, serving as an integrative indicator of disease activity.
  The numbers 0 and 10 are written at both ends of a 10 cm line. 0 = very much worse 10 = much better The PGA level increases from 0 to 10. The patient is asked to indicate which point on this chart is most appropriate for his/her situation. The location marked by the patient will be evaluated by measuring its distance from point 0.

CONTACTS AND LOCATIONS:
Overall Officials: Birkan Sonel Tur, Prof, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corti MC, Rigon C. Epidemiology of osteoarthritis: prevalence, risk factors and functional impact. Aging Clin Exp Res. 2003 Oct;15(5):359-63. doi: 10.1007/BF03327356. PMID 14703001
- [Background] Driban JB, Harkey MS, Barbe MF, Ward RJ, MacKay JW, Davis JE, Lu B, Price LL, Eaton CB, Lo GH, McAlindon TE. Risk factors and the natural history of accelerated knee osteoarthritis: a narrative review. BMC Musculoskelet Disord. 2020 May 29;21(1):332. doi: 10.1186/s12891-020-03367-2. PMID 32471412
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Nelson AE, Allen KD, Golightly YM, Goode AP, Jordan JM. A systematic review of recommendations and guidelines for the management of osteoarthritis: The chronic osteoarthritis management initiative of the U.S. bone and joint initiative. Semin Arthritis Rheum. 2014 Jun;43(6):701-12. doi: 10.1016/j.semarthrit.2013.11.012. Epub 2013 Dec 4. PMID 24387819
- [Background] Haupt G. Use of extracorporeal shock waves in the treatment of pseudarthrosis, tendinopathy and other orthopedic diseases. J Urol. 1997 Jul;158(1):4-11. doi: 10.1097/00005392-199707000-00003. PMID 9186313
- [Background] Sems A, Dimeff R, Iannotti JP. Extracorporeal shock wave therapy in the treatment of chronic tendinopathies. J Am Acad Orthop Surg. 2006 Apr;14(4):195-204. doi: 10.5435/00124635-200604000-00001. PMID 16585361
- [Background] Wang CJ. Extracorporeal shockwave therapy in musculoskeletal disorders. J Orthop Surg Res. 2012 Mar 20;7:11. doi: 10.1186/1749-799X-7-11. PMID 22433113
- [Background] Wang CJ, Sun YC, Siu KK, Wu CT. Extracorporeal shockwave therapy shows site-specific effects in osteoarthritis of the knee in rats. J Surg Res. 2013 Aug;183(2):612-9. doi: 10.1016/j.jss.2013.02.006. Epub 2013 Feb 26. PMID 23472862
- [Background] Zhao Z, Jing R, Shi Z, Zhao B, Ai Q, Xing G. Efficacy of extracorporeal shockwave therapy for knee osteoarthritis: a randomized controlled trial. J Surg Res. 2013 Dec;185(2):661-6. doi: 10.1016/j.jss.2013.07.004. Epub 2013 Jul 30. PMID 23953895
- [Background] Lee JK, Lee BY, Shin WY, An MJ, Jung KI, Yoon SR. Effect of Extracorporeal Shockwave Therapy Versus Intra-articular Injections of Hyaluronic Acid for the Treatment of Knee Osteoarthritis. Ann Rehabil Med. 2017 Oct;41(5):828-835. doi: 10.5535/arm.2017.41.5.828. Epub 2017 Oct 31. PMID 29201822
- [Background] Zhong Z, Liu B, Liu G, Chen J, Li Y, Chen J, Liu X, Hu Y. A Randomized Controlled Trial on the Effects of Low-Dose Extracorporeal Shockwave Therapy in Patients With Knee Osteoarthritis. Arch Phys Med Rehabil. 2019 Sep;100(9):1695-1702. doi: 10.1016/j.apmr.2019.04.020. Epub 2019 Jun 10. PMID 31194946